CLINICAL TRIAL: NCT05297942
Title: Effect of Expansion of Abbreviations and Acronyms on Patient Comprehension of Their Health Records: A Randomized Clinical Trial
Brief Title: Expansion of Abbreviations and Acronyms for Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1804019182
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: Abbreviations; Acronyms; Personal Health Records; Patient Portals; Consumer Health Informatics; Patient Access to Records
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: Masking not possible due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Expansion) Arm (Experimental): Expansion of abbreviations and acronyms
  Interventions: Other: Expansion of Abbreviations and Acronyms
- Control (Abbreviation) Arm (No Intervention): No expansion of abbreviations and acronyms

INTERVENTIONS:
Other: Expansion of Abbreviations and Acronyms — Expansion of Abbreviations and Acronyms
  Arms: Intervention (Expansion) Arm

SUMMARY:
This is a prospective, two-arm, parallel, individually randomized controlled trial to estimate the effect of expansion on patient comprehension (primary outcome) of abbreviations and acronyms in their health records. English-speaking adult patients with diagnosed heart failure who receive primary care at three urban hospitals in New York City will be considered. The investigators hypothesize that expansion will significantly increase patient comprehension of abbreviations and acronyms in the health record.

DETAILED DESCRIPTION:
Importance: In 2020, an estimated 100 million Americans accessed their own health records online. That number likely increased beginning April 2021, when U.S. federal rules implemented the 21st Century Cures Act requiring electronic health information to be made freely accessible. Medical abbreviations and acronyms may limit patient understanding of health records. Automated expansion is one potential solution, however, the magnitude of its effect on patient comprehension has not been estimated.

Objective: To estimate the effect of expansion on patient comprehension of abbreviations and acronyms in their health records.

Design: Prospective, two-arm, parallel, individually randomized controlled trial.

Participants: Patients who receive primary care at one of three urban hospitals. A purposive sample representative on age, gender, and race will be enrolled between February 2020 and August 2021. To isolate the main effect, the investigators will include only English-speaking adult patients with diagnosed heart failure.

Intervention: Participants will be randomized to receive clinical text with abbreviations (control group, n=30) or with expansions (intervention group, n=30). The abbreviations and expansions included "hrs" (hours), "MD" (medical doctor), "BP" (blood pressure), "ED" (emergency department), "yo" (year old), "pt" (patient), "HF" (heart failure), "hx" (history), "HTN" (hypertension), "MI" (myocardial infarction).

ELIGIBILITY:
Inclusion Criteria:

* Adult (21 years or older)
* Confirmed diagnosis of heart failure
* Able to read and speak English
* Willing and able to provide informed consent
* Receives primary care from participating provider

Exclusion Criteria:

* Healthcare professional (MD, DO, RN, etc.)
* No telephone number or email address
* Severe cognitive impairment or clinical diagnosis of dementia
* Major psychiatric illness, including active psychosis
* Other illness that would preclude participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Overall comprehension | Day 1, at the time of the intervention administration
  count of the total number of abbreviated or expanded terms comprehended by the each participant

CONTACTS AND LOCATIONS:
Overall Officials: Ruth M Masterson Creber, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed study will generate data on comprehension from 60 recently hospitalized patients with advanced heart failure. The final locked dataset will be shared with other investigators or healthcare organizations upon request and without cost. Before the request is fulfilled, the investigator or organization must sign a data-sharing agreement to demonstrate and provide for: (1) a commitment to using the information only for research or clinical purposes and not to identify any individual participant, (2) a commitment to securing the information using appropriate computer technology, (3) a commitment to not share the information outside the immediate research or clinical setting, and (4) a commitment to erasing the data after the analyses are completed.
Supporting Information: Study Protocol, SAP
Time Frame: The trial protocol and statistical analysis plan will be made available upon publication
Access Criteria: Public

REFERENCES:
- [Result] Grossman Liu L, Russell D, Reading Turchioe M, Myers AC, Vawdrey DK, Masterson Creber RM. Effect of Expansion of Abbreviations and Acronyms on Patient Comprehension of Their Health Records: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2212320. doi: 10.1001/jamanetworkopen.2022.12320. PMID 35560053